CLINICAL TRIAL: NCT01626742
Title: A Randomized Double Blinded Controlled Trial of an Oral Nutritional Supplement Containing AN 777 in Older Hospitalized Patients
Brief Title: A Trial of an Oral Nutritional Supplement in Older Hospitalized Patients - NOURISH Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BL01
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Hospitalized Elderly

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ready to drink flavored beverage (Placebo Comparator)
  Interventions: Other: Ready to Drink Flavored Beverage
- Ready to drink flavored beverage w/ AN 777 (Experimental)
  Interventions: Other: Ready to drink flavored beverage w/ AN 777

INTERVENTIONS:
Other: Ready to Drink Flavored Beverage — 2 servings a day
  Arms: Ready to drink flavored beverage
Other: Ready to drink flavored beverage w/ AN 777 — 2 servings a day
  Arms: Ready to drink flavored beverage w/ AN 777

SUMMARY:
Evaluate effects of an oral nutritional supplement on healthcare outcomes in older hospitalized adults. Also referred to as the NOURISH Study - Nutrition effect On Unplanned Readmissions and Survival in Hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 65 years of age.
2. Admitted to hospital with diagnosis of heart failure, acute myocardial infarction, pneumonia, or chronic obstructive pulmonary disease.
3. Subjective Global Assessment rating of B or C.
4. Length of hospital stay anticipated to be > 3 days and < 12 days
5. Able to consume foods and beverages orally.
6. Functionally ambulatory during the 30 days prior to admission.

Exclusion Criteria:

1. Uncontrolled hypertension
2. Diagnosis of diabetes
3. Current active cancer or recently treated cancer
4. Impaired renal function
5. Liver failure, acute Hepatitis, or hepatic encephalopathy
6. Active tuberculosis.
7. HIV
8. Disorder of gastrointestinal tract
9. Autoimmune disorder
10. Intubation, and/or tube or parenteral feeding.
11. Severe dementia or delirium, brain metastases, eating disorder, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
12. Allergy or intolerance to any of the ingredients in the study products.
13. Body mass index of ≥ 40 kg/m2.
14. Resident in a nursing home or other residential facility.
15. Planned surgery during course of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 652 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Return to hospital or death | 90 days

SECONDARY OUTCOMES:
Return to hospital or death | 30 and 60 days
Hospital Days | 90 days
Activities of Daily Living | 90 days
  Katz Activities of Daily Living at entry and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Luo, MD, PhD, Study Chair — Abbott Nutrition; Jeffrey Nelson, PhD, Study Chair — Abbott Nutrition
Locations (118):
- United States (114):
  - Auburn University, Auburn, Alabama
  - Birmingham Heart Clinic, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - HealthScan Research, Montgomery, Alabama
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - UCSF Fresno, Fresno, California
  - St. Jude Medical Center, Fullerton, California
  - Glendale Adventist Medical Center, Glendale, California
  - eStudySite, La Mesa, La Mesa, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Novo Research dba FCPP Research, Modesto, California
  - eStudySite, Oceanside, Oceanside, California
  - Pulmonary Consultant & Primary Physicians Medical Group, Orange, California
  - Los Angeles Biomedical Research Institution, Torrance, California
  - Aurora Denver Cardiology Associates, PC, Aurora, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - UConn Health Center, Farmington, Connecticut
  - ZASA Clinical Research, Atlantis, Florida
  - Visions Clinical Research, LLC, Boynton Beach, Florida
  - Pulmonary and Sleep of Tampa Bay, Brandon, Florida
  - Morton Plant Mease HealthCare, Clearwater, Florida
  - Seidman Clinical Trials, Delray Beach, Florida
  - Broward Health - Broward General Medical Center, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - In Vivo Clinical Research, Hialeah, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - The Cardiovascular Center, P.A., Lake Mary, Florida
  - Watson Clinic Center for Research, Inc., Lakeland, Florida
  - Largo Medical Center, Largo, Florida
  - Panama Clinical Research Associates, Lynn Haven, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Cuervo Clinical Research Group, Inc, Miami, Florida
  - Health & Life Research Solutions Inc., Miami, Florida
  - Ocala Research Institute, Inc., Ocala, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Regenerate Clinical Trials, South Miami, Florida
  - Advanced Clinical Research Group, Stuart, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Emory University, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Atlanta Institute for Medical Research, Decatur, Georgia
  - Kootenai Heart Clinics, LLC, Coeur d'Alene, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Edward Hines VA Hospital, Hines, Illinois
  - St Vincent Medical Group, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - King's Daughters Medical Center, Kentucky Heart Foundation , Inc., Ashland, Kentucky
  - Research Concierge, LLC, Hartford, Kentucky
  - Kentucky Lung Clinic, Hazard, Kentucky
  - Jewish Hospital & St Mary's Healthcare, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Louisiana State University Health Science Center, Shreveport, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MedStar Health Research Institute - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Activmed Practices & Research, Inc, Methuen, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - McLaren-Flint Research Institute, Flint, Michigan
  - St John Hospital & Medical Center, Grosse Pointe Woods, Michigan
  - Bronson Healthcare Group, Kalamazoo, Michigan
  - Crittenton Hospital Medical Center, Rochester Hills, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - HealthEast St Joseph's Hospital, Saint Paul, Minnesota
  - David M Headley, Port Gibson, Mississippi
  - St Anthony's Medical Center, St Louis, Missouri
  - Alegent Creighton Health Heart & Vascular Specialists, Omaha, Nebraska
  - Creighton University, Omaha, Nebraska
  - eStudySite, Las Vegas, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Hunterdon Cardiovascular Associates, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Virtua Medical Group, Moorestown, New Jersey
  - Associated Cardiovascular Consultants of Lourdes, Voorhees Township, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Erie County Medical Center, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Mission Hospital, Asheville, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Novant Clinical Research Institute, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - The Carl and Edyth Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - North Ohio Research, Elyria, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Physician Specialists of Northern Lancaster County Medical Group, Ephrata, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Inc., Sayre, Pennsylvania
  - Grand View Hospital Clinical Research, Sellersville, Pennsylvania
  - The Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Inc., Wormleysburg, Pennsylvania
  - PMG research of Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Senior Primary Care Practice, Columbia, South Carolina
  - Sanford Clinic Family Medicine, Sioux Falls, South Dakota
  - STHS Heart, LLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas A&M University, College Station, Texas
  - Advanced Clinical Research Associates, Plano, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Sonterra Clinical Research, San Antonio, Texas
  - Tanner Clinic, Layton, Utah
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Carilion Medical Center Geriatrics, Roanoke, Virginia
  - Salem VA Medical Center, Salem, Virginia
  - The Hope Heart Institute, Bellevue, Washington
- Puerto Rico (4):
  - San Juan Bautista School of Medicine, Caguas
  - Western Cardiovascular Surgery of Puerto Rico, Mayagüez
  - Research and Cardiovascular Corp, Ponce
  - VA Caribbean Healthcare System, San Juan

REFERENCES:
- [Derived] Baggs GE, Middleton C, Nelson JL, Pereira SL, Hegazi RM, Matarese L, Matheson E, Ziegler TR, Tappenden KA, Deutz N. Impact of a specialized oral nutritional supplement on quality of life in older adults following hospitalization: Post-hoc analysis of the NOURISH trial. Clin Nutr. 2023 Nov;42(11):2116-2123. doi: 10.1016/j.clnu.2023.09.004. Epub 2023 Sep 9. PMID 37757502
- [Derived] Matheson EM, Nelson JL, Baggs GE, Luo M, Deutz NE. Specialized oral nutritional supplement (ONS) improves handgrip strength in hospitalized, malnourished older patients with cardiovascular and pulmonary disease: A randomized clinical trial. Clin Nutr. 2021 Mar;40(3):844-849. doi: 10.1016/j.clnu.2020.08.035. Epub 2020 Sep 5. PMID 32943241
- [Derived] Deutz NE, Matheson EM, Matarese LE, Luo M, Baggs GE, Nelson JL, Hegazi RA, Tappenden KA, Ziegler TR; NOURISH Study Group. Readmission and mortality in malnourished, older, hospitalized adults treated with a specialized oral nutritional supplement: A randomized clinical trial. Clin Nutr. 2016 Feb;35(1):18-26. doi: 10.1016/j.clnu.2015.12.010. Epub 2016 Jan 18. PMID 26797412